CLINICAL TRIAL: NCT03146065
Title: A Phase 1, Randomized, Double Blind, Sponsor-open, Placebo-controlled, First-in-human Trial To Evaluate The Safety, Tolerability, And Pharmacokinetics Of Pf-06730512 After Single And Multiple Ascending Intravenous Infusion Or Subcutaneous Administration To Healthy Adult Subjects And An Open-label Evaluation In Healthy Japanese Subjects
Brief Title: Evaluation Of Safety, Tolerability And Pharmacokinetics Of Single And Multiple Doses Of PF-06730512
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Basic Science
Other Study IDs: C0221001; 2016-004493-18 (EudraCT Number); FIH SAD/MAD (Other: Alias Study Number)
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Healthy
MeSH Terms: interventions — PF-06730512

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PF-06730512 (Experimental): Study Drug being used in the study
  Interventions: Biological: PF-06730512
- Placebo (Placebo Comparator): Placebo for IV/SC administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: PF-06730512 — Comparison of different dosages of PF-06730512 to Placebo
  Arms: PF-06730512
Drug: Placebo — Comparison of Placebo to different doses of PF-06730512
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety, tolerability and pharmacokinetics of escalating single and multiple intravenous (IV) infusions and subcutaneous (SC) injections of PF-06730512 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects of nonchildbearing potential and/or male subjects who, at the time of screening, are between the ages of 18 and 55 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure (BP) and pulse rate (PR) measurement, 12-lead electrocardiogram (ECG), or clinical laboratory tests.
* Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).

Exclusion Criteria:

- History of allergic reactions to diagnostic or therapeutic protein. History of recurrent infections or active infection within 28 days of screening.

Exposure to live vaccines within 28 days of screening.

- History of human immunodeficiency virus (HIV), hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen (HepBsAg), hepatitis B core antibody (HepBcAb), or hepatitis C antibody (HCVAb). As an exception, a positive hepatitis B surface antibody (HBsAb) finding as a result of subject vaccination is permissible.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2018-05-03 (Actual); Study Completion 2018-05-03 (Actual)

PRIMARY OUTCOMES:
Number of Subjects With Treatment Emergent Treatment-Related Adverse Event(s) | Dosing through approximately Day 71 (single dose) or Day 113 (multiple dose)
  Number of Subjects With Treatment Emergent Treatment-Related Adverse Event(s)
Number of subjects with injection site reaction(s) | Dosing through approximately Day 71 (single dose) or Day 113 (multiple dose)
  Number of subjects with injection site reaction(s)
Number of subjects with laboratory test findings of potential clinical importance | Dosing through approximately Day 71 (single dose) or Day 113 (multiple dose)
  Number of subjects with laboratory test findings of potential clinical importance
Number of subjects with vital signs findings of potential clinical importance | Dosing through approximately Day 71 (single dose) or Day 113 (multiple dose)
  Number of subjects with vital signs findings of potential clinical importance
Number of subjects with ECG findings of potential clinical importance | Dosing through approximately Day 71 (single dose) or Day 113 (multiple dose)
  Number of subjects with ECG findings of potential clinical importance

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of PF-06730512 | Day 1 to approximately Day 71 (single dose) or Day 113 (multiple dose)
  Maximum Observed Plasma Concentration (Cmax) of PF-06730512
Time to Reach Maximum Observed Concentration (Tmax) of PF-06730512 | Day 1 to approximately Day 71 (single dose) or Day 113 (multiple dose)
  Time to Reach Maximum Observed Concentration (Tmax) of PF-06730512
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of PF-06730512 | Day 1 to approximately Day 71 (single dose) or Day 113 (multiple dose)
  Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of PF-06730512
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0- infinity)] of PF-06730512, as permitted | Day 1 to approximately Day 71 (single dose) or Day 113 (multiple dose)
  Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0- infinity)] of PF-06730512, as permitted
Clearance (CL) or Apparent Clearance (CL/F) of PF-06730512, as permitted | Day 1 to approximately Day 71 (single dose) or Day 113 (multiple dose)
  Clearance (CL) or Apparent Clearance (CL/F) of PF-06730512, as permitted
Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) of PF-06730512 | Day 1 to approximately Day 113
  Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) of PF-06730512
Apparent Volume of Distribution of PF-06730512, as permitted | Day 1 to approximately Day 71 (single dose) or Day 113 (multiple dose)
  Apparent Volume of Distribution of PF-06730512, as permitted
Terminal half-life, as permitted | Day 1 to approximately Day 71 (single dose) or Day 113 (multiple dose)
  Terminal half-life, as permitted
Accumulation ratio (Rac), as permitted | Day 1 to approximately Day 113
  Accumulation ratio (Rac), as permitted
Minimum observed concentration during the dosing interval (Cmin) | Day 1 to approximately Day 113
  Minimum observed concentration during the dosing interval (Cmin)
Incidence of the development of anti-drug antibody (ADA) and neutralizing antibody (NAb) | Day 1 to approximately Day 71 (single dose) or Day 113 (multiple dose)
  Incidence of the development of anti-drug antibody (ADA) and neutralizing antibody (NAb)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
Information relating to our policy on data sharing and the process for requesting data can be found at the following link: http://www.pfizer.com/research/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Lim CN, Kantaridis C, Huyghe I, Gorman D, Berasi S, Sonnenberg GE. A Phase 1 first-in-human study of the safety, tolerability, and pharmacokinetics of the ROBO2 fusion protein PF-06730512 in healthy participants. Pharmacol Res Perspect. 2021 Aug;9(4):e00813. doi: 10.1002/prp2.813. PMID 34369667
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=C0221001&StudyName=A+Phase+1%2C+Randomized%2C+Double+Blind%2C+Sponsor-open%2C+Placebo+Controlled%2C+First-in-human+Trial+To+Evaluate+The+Safety%2C+Tolerability%2C+And+Pharmacokinetics+Of+Pf+06730512+After+Single+And+Multiple+Ascending+Intravenous+Infusion+Or+Subcutaneous+Administration+To+Healthy+Adult+Subjects+And+An+Open-label+Evaluation+In+Healthy+Japanese+Subjects
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=C0221001&StudyName=A+Phase+1%2C+Randomized%2C+Double+Blind%2C+Sponsor-open%2C+Placebo-controlled%2C+First-in-human+Trial+To+Evaluate+The+Safety%2C+Tolerability%2C+And+Pharmacokinetics+Of+Pf-06730512+After+Single+And+Multiple+Ascending+Intravenous+Infusion+Or+Subcutaneous+Administration+To+Healthy+Adult+Subjects+And+An+Open-label+Evaluation+In+Healthy+Japanese+Subjects